CLINICAL TRIAL: NCT04806594
Title: Open Label, Uncontrolled Clinical Investigation on the Safety and Clinical Performance of Papix Acne Scar in the Prevention and Improvement of Scars and Lesions Associated With Acne
Brief Title: Clinical Investigation on the Safety and Clinical Performance of Papix Acne Scar.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Relife S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReGl/19/PAS-Acn/001
Record Dates: First submitted 2020-11-13; First posted 2021-03-19 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Acne; Scars
Keywords: cream; mild moderate acne; Papix; Papix acne scar; acne treatment
MeSH Terms: conditions — Acne Vulgaris; Cicatrix

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, uncontrolled, single arm, post-market clinical follow-up study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Papix acne scar (Experimental): Papix acne scar gel for 8 consecutive weeks, 2 times per day
  Interventions: Device: Papix acne scar

INTERVENTIONS:
Device: Papix acne scar — PapiX acne scar, class IIa medical device, gel for acne scar. to be applied 2 times per day during the 8 weeks of study duration

SUMMARY:
The scope of this open label clinical trial is to evaluate and confirm the performance of Papix acne scar in the prevention and improvement of acne scars in subject suffering for mild to moderate acne. The product will be applied for 8 consecutive weeks and 3 clinical follow up visits will be performed.

DETAILED DESCRIPTION:
The scope of this open label clinical trial is to evaluate and confirm the performance of Papix acne scar in the prevention and improvement of acne scars in subject suffering for mild to moderate acne. The product will be applied for 8 consecutive weeks, 2 times per day into the face.

The dermatologist will perform 3 clinical follow up visits to assess the efficacy and safety of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's or parents or guardian (depending on the age of the subject) written informed consent obtained prior to any study-related procedures;
2. Male or female subjects aged ≥ 12 years of any race;
3. Subjects with any Fitzpatrick skin phototype;
4. Subjects with clinical diagnosis of mild to moderate acne vulgaris (IGA score 2 or 3) on the face;
5. Presence of acne scars (all types included), of grade mild or moderate according to SGA;
6. Subjects with cooperative attitude, able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and able to comply with the requirements of the entire investigation (including ability to attend the planned visits according to the time limits), based on Investigator's judgement.

Exclusion Criteria:

1. Pregnant women
2. Severe acne at inclusion or any acne requiring systemic treatment;
3. Presence of facial warts or fungal infections;
4. Active dermatitis on the face, rosacea, active herpes simplex;
5. Keloids presence in the area to be treated or keloids development during the treatment period;
6. History of radiation or skin tumors in the/close to the area to be treated in the past 5 years;
7. Laser ablative procedures within the last month;
8. Chemical peels within the last 6 months;
9. Use of topical treatments like antibiotics, corticosteroids, benzoyl peroxide, azelaic acid, hydroxy acids and other antinflammatory drugs within 2 weeks;
10. Use of topical retinoids within 4 weeks;
11. Use of systemic corticosteroids or antibiotics in the previous 30 days;
12. Use of systemic spironolactone/drospirenone or immunomodulators in the previous 3 months;
13. Use of oral retinoids or cyproterone acetate/chlormadinone acetate in the previous 6 months;
14. Use of scrub, alpha hydroxy acid (AHA), skin irritant products in the 2 days before study treatment start;
15. Subjects with any other clinically significant or unstable concurrent disease or skin condition or general condition that, in the Investigator's opinion, might interfere with the study evaluations;
16. Allergy, sensitivity or intolerance to the components of the investigational device formulations ingredients;
17. Concomitant or previous participation in other interventional clinical study in the past 3 months;
18. Subjects planning sun exposure or tanning booths or UV sources throughout the course of the study. In case of sun exposure this shall be limited and a protection cream (SPF 50+) shall be applied.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Parodi, Principal Investigator — Ospedale Policlinico San Martino
Locations (1):
- Ospedale San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 40 subjects were enrolled in the study and 39 of them started the treatment, 9 male (23.1%) and 30 females (76.9%). The global range was between 12 and 65 years. Overall, three subjects interrupted prematurely the study (one of them never started the treatment and two withdrew during the study).
Groups:
- PAPIX ACNE SCAR, Topically Applied Twice a Day for 8 Weeks.: Papix acne scar gel for 8 consecutive weeks, 2 times per day
  PAPIX ACNE SCAR was topically applied twice a day for 8 weeks, 2 FTU (finger-tip units) in the morning and in 2 FTU the evening before bedtime, on the face, and massaged gently into the skin until absorbed.
Period: Overall Study
Arm/Group | PAPIX ACNE SCAR, Topically Applied Twice a Day for 8 Weeks.
Started | 40
Completed | 37
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Did never apply the study product and did not attend following visits. | 1

BASELINE CHARACTERISTICS:
Population: 39 partecipants are the FAS
Groups:
- PAPIX ACNE SCAR, Topically Applied Twice a Day for 8 Weeks.: Patients will be instructed to use PAPIX ACNE SCAR applied twice a day, in the morning and in the evening before bedtime, and massaged gently into the skin until absorbed. PAPIX ACNE SCAR shall be applied only on the lesions, where possible. The treatment duration will be of 8 weeks
Arm/Group | PAPIX ACNE SCAR, Topically Applied Twice a Day for 8 Weeks.
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants] — Population: A total of 40 subjects were enrolled in the study and 39 of them started the treatment, 9 male (23.1%) and 30 females (76.9%). The global range was between 12 and 65 years. Overall, three subjects interrupted prematurely the study (one of them never started the treatment and two withdrew during the study).
  Participants
    <=18 years | 11
    Between 18 and 65 years | 28
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — total of 40 subjects were enrolled in the study and 39 of them started the treatment, 9 male (23.1%) and 30 females (76.9%).
  Participants
    Female | 30
    Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — The clinical investigation involved two clinical sites, the coordinating site (site 01) IRCCS San Martino - Genova - P.I. Prof. Aurora Parodi and the satellite site (site 02) IRCCS Gaslini - Genova - P.I. Prof. Corrado Ocella. Both clinical sites were allocated in Liguria (Italy)
  Participants
    Italy | 39
Subjects had clinical diagnosis of mild to moderate acne vulgaris on the face [Count of Participants; unit: Participants] — (IGA score 2 or 3)
  Participants | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Partecipants With Improvement of Acne Scars and Marks and Without New Acne Scars After 4 Weeks
Description: The primary endpoint will be the proportion of subjects with acne scars and marks improved with respect to baseline and, at the same time, without any new facial acne scars after 4 weeks of treatment (treatment success). The improvement of acne scars and marks will be assessed as the change of at least one grade in the qualitative Scar Global Assessment (SGA) by Goodman and Baron between baseline and Week 4. The number of new acne scars will be assessed by count and comparison with baseline.
Time Frame: four weeks of treatment
Population: PPAS population: Per-Protocol analysis set (PPAS): all patients of the FAS who also meet all inclusion/exclusion criteria and who do not have any major protocol deviation (i.e. wrong inclusion, use of forbidden concomitant medications, etc.).
Measure: Number; unit: participants
Groups:
- No. 39 Subjects, Male or Female, Aged ≥ 12 Years, of Any Race, With Any Fitzpatrick Skin Phototype: Papix acne scar gel for 8 consecutive weeks, 2 times per day
  Papix acne scar: PapiX acne scar, class IIa medical device, gel for acne scar. to be applied 2 times per day during the 8 weeks of study duration
Arm/Group | No. 39 Subjects, Male or Female, Aged ≥ 12 Years, of Any Race, With Any Fitzpatrick Skin Phototype
Number analyzed (Participants) | 39
participants | 5

2. Secondary Outcome: Number of Partecipants With Improvement of Acne Scars and Marks and Without New Acne Scars After Treatment
Description: Indicate the proportion of subjects with improved acne scars and marks with respect to baseline and, at the same time, without any new facial acne scars after 2 and 8 weeks of treatment. The improvement of acne scars and marks will be assessed as the change in the qualitative Scar Global Assessment (SGA) questionnaire
Time Frame: two weeks of treatment and 8 weeks of treatment, week 8 reported
Population: Per-Protocol analysis set (PPAS): all patients of the FAS who also meet all inclusion/exclusion criteria and who do not have any major protocol deviation (i.e. wrong inclusion, use of forbidden concomitant medications, etc.).
Measure: Count of Participants; unit: Participants
Groups:
- Proportion of Subjects With Improved Acne Scars and Marks at Week 2 and 8 of Treatment: To evaluate the performance of PAPIX ACNE SCAR in the prevention and improvement of acne scars after 2 and 8 weeks of treatment. This endpoint will be assessed as the proportion of subjects with improved acne scars and marks with respect to baseline and, at the same time, without any new facial acne scars after 2 and 8 weeks of treatment. The improvement of acne scars and marks will be assessed as the change in the qualitative Scar Global Assessment (SGA) between baseline and Week 2 and 8. The number of acne scars, to identify any new scars, will be assessed through the scars count and comparison with baseline.
Arm/Group | Proportion of Subjects With Improved Acne Scars and Marks at Week 2 and 8 of Treatment
Number analyzed (Participants) | 37
Participants | 22

3. Secondary Outcome: Number of Partecipants With Improvement of Acne Scars and Marks and Without New Acne Scars After Treatment
Description: Proportion of subjects at week 2, 4 and 8 of treatment, without any new facial acne lesions with respect to baseline (Visit 1).
Time Frame: assested at two weeks, 4 weeks and 8 weeks, week 8 reported
Measure: Count of Participants; unit: Participants
Groups:
- New Facial Acne Lesions With Respect to Baseline at Week 2, 4 and 8 of Treatment: To evaluate the performance of PAPIX ACNE SCAR in the prevention of acne lesions after 2, 4 and 8 weeks of treatment. The number of acne lesions, to identify any new lesions, will be assessed through the lesions count and comparison with baseline.
Arm/Group | New Facial Acne Lesions With Respect to Baseline at Week 2, 4 and 8 of Treatment
Number analyzed (Participants) | 37
Participants | 33

4. Secondary Outcome: Acne Investigator Global Assessment (IGA) Scores
Description: To evaluate acne severity after 2 weeks (visit 2), 4weeks (visit 3) and 8 weeks (visit 4) of treatment, through the Investigator Global Assessment.
  Acne Investigator Global Assessment (IGA). Five different grades were used to define the acne severity: 0 Clear, 1 Almost Clear, 2 Mild, 3 Moderate, 4 Severe;
Time Frame: assested at two weeks (visit 2), 4 weeks (visit 3) and 8 weeks (visit 4)
Population: Due to protocol deviation some subjects were not included in all outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Change From Baseline (Visit 1) to Each Time Point (Visit 2, 3 and 4) in the Acne Severity: To evaluate the improvement in acne severity after 2 weeks (visit 2), 4weeks (visit 3) and 8 weeks (visit 4) of treatment, through the Investigator Global Assessment, ranging from 0 (clear; clear skin with no lesions) to 4 (severe; many inflammatory and non- inflammatory lesions).
Arm/Group | Change From Baseline (Visit 1) to Each Time Point (Visit 2, 3 and 4) in the Acne Severity
Number analyzed (Participants) | 39
score on a scale
  Change of IGA from baseline to Visit 2 (2 weeks) | -0.86 (0.28)
  Change of IGA from baseline to Visit 3 (4 weeks): number analyzed (Participants) | 35
  Change of IGA from baseline to Visit 3 (4 weeks) | -0.26 (0.51)
  Change of IGA from baseline to Visit 4 (8 weeks): number analyzed (Participants) | 37
  Change of IGA from baseline to Visit 4 (8 weeks) | -0.86 (0.67)

5. Secondary Outcome: Change of Skin Roughness
Description: To evaluate the improvement of the skin roughness after 2, 4 and 8 weeks of treatment.through the Investigator Global Assessment Acne Investigator Global Assessment (IGA)
Time Frame: assested at two weeks, 4 weeks (visit 3) and 8 weeks (visit 4)
Population: Due to protocol deviation some subjects were not included in all outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Change From Baseline (Visit 1) to Each Following Time Point in the Skin Roughness: To evaluate the improvement of the skin roughness on a 4-point scale from 0 (none; very smooth) to 3 (severe; very rough) after 2, 4 and 8 weeks of treatment.
Arm/Group | Change From Baseline (Visit 1) to Each Following Time Point in the Skin Roughness
Number analyzed (Participants) | 39
score on a scale
  Change of skin roughness assessment from baseline to Visit 2 (2 weeks) | -0.38 (0.35)
  Change of skin roughness assessment from baseline to Visit 3 (4 weeks): number analyzed (Participants) | 35
  Change of skin roughness assessment from baseline to Visit 3 (4 weeks) | -0.11 (0.40)
  Change of skin roughness assessment from baseline to Visit 4 ( 8 weeks): number analyzed (Participants) | 37
  Change of skin roughness assessment from baseline to Visit 4 ( 8 weeks) | -0.38 (0.64)

6. Secondary Outcome: Number of Partecipants With Skin Texture Improvement
Description: To evaluate the change in skin texture after 2, 4 and 8 weeks of treatment, through the Investigator Global Assessment. Acne Investigator Global Assessment (IGA).
Time Frame: assested at two weeks, 4 weeks and 8 weeks, week 8 reported
Measure: Count of Participants; unit: Participants
Groups:
- Change From Baseline (Visit 1) to Each Time Point (Visit 2, 3 and 4) in the Skin Texture: Change from baseline (Visit 1) to each time point (Visit 2, 3 and 4) in the skin texture on a 6-point scale from 0 (worse) to 5 (complete improvement).
Arm/Group | Change From Baseline (Visit 1) to Each Time Point (Visit 2, 3 and 4) in the Skin Texture
Number analyzed (Participants) | 37
Participants | 16

7. Secondary Outcome: Number of Partecipants Compliant to Treatment
Description: To evaluate the subject's adherence to treatment by the product accountability.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Subject's Adherence to Treatment: The number of applications will be self-reported by the subject to assess adherence to treatment.
Arm/Group | Subject's Adherence to Treatment
Number analyzed (Participants) | 37
Participants | 37

8. Secondary Outcome: Subject and Investigator Global Evaluation of Performance
Description: To evaluate the subject's and Investigator's global evaluation of satisfaction with regards to the performance of PAPIX ACNE SCAR through a specific questionnaire.
Time Frame: 8 weeks of treatment ( visit 4)
Measure: Count of Participants; unit: Participants
Groups:
- Subject's and Investigator's Global Evaluation of Satisfaction: Subject's and Investigator's global evaluation on performance of the study product at the end of the study (Visit 4) by means of a 7-items scale.
Arm/Group | Subject's and Investigator's Global Evaluation of Satisfaction
Number analyzed (Participants) | 37
Participants
  Subject's global evaluation of performance: Very much improved | 7
  Subject's global evaluation of performance: Improved | 13
  Subject's global evaluation of performance: Minimally improved | 11
  Subject's global evaluation of performance: No change | 4
  Subject's global evaluation of performance: Worse | 2
  Investigator's global evaluation of performance: Very much improved | 1
  Investigator's global evaluation of performance: Improved | 19
  Investigator's global evaluation of performance: Minimally improved | 8
  Investigator's global evaluation of performance: No change | 7
  Investigator's global evaluation of performance: Worse | 2

9. Secondary Outcome: Treatment Acceptability
Description: To evaluate the subject's overall acceptability of the treatment through a specific questionnaire.
Time Frame: 8 weeks of treatment ( visit 4)
Measure: Count of Participants; unit: Participants
Groups:
- Subject's Overall Acceptability of the Treatment,: Subject's overall acceptability of the treatment at the end of the study (Visit 4) by means of a 5-item scale.
Arm/Group | Subject's Overall Acceptability of the Treatment,
Number analyzed (Participants) | 37
Participants
  Very much satisfied | 7
  Satisfied | 19
  Neither satisfied nor dissatisfied | 8
  Dissatisfied | 2
  Very much dissatisfied | 1

10. Other Pre Specified Outcome: Number of Partecipants With Adverse Events
Description: To evaluate the local and general tolerability of PAPIX ACNE SCAR.
Time Frame: two weeks, 4 weeks and 8 weeks of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Adverce Events: To evaluate the local and general tolerability of PAPIX ACNE SCAR. Adverse events and adverse reactions will be recorded and evaluated.
Arm/Group | Adverce Events
Number analyzed (Participants) | 39
Participants | 1

ADVERSE EVENTS:
Time Frame: All subjects enrolled were treated with PAPIX ACNE SCARS for 8 weeks
Description: Only one adverse event was registered during the study. The event was not related to the study treatment (mild foot contusion).
Groups:
- Safety Population): To evaluate the local and general tolerability of PAPIX ACNE SCAR. Adverse events and adverse reactions were recorded and evaluated.
Arm/Group | Safety Population)
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population) (N=40)
mild foot contusion). (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04806594/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT04806594/SAP_001.pdf